CLINICAL TRIAL: NCT00207467
Title: Prospective Study for Cost-Effectiveness Strategies to Improve Partner Notification: Female Trichomonas and Male Urethritis Studies
Brief Title: Study to Improve Partner Services for STD Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3196; CA# R30/CCR619143-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Trichomonas Vaginalis; Urethritis
Keywords: patient-delivered partner treatment; partner referral; sexually transmitted diseases
MeSH Terms: conditions — Urethritis; Sexually Transmitted Diseases

INTERVENTIONS:
Behavioral: Patient-delivered partner treatment
Behavioral: Booklet-enhanced partner referral

SUMMARY:
The goal of this study was to examine the efficacy of patient-delivered partner treatment (PDPT) compared to standard partner referral (PR) and booklet enhanced partner referral (BEPR).

DETAILED DESCRIPTION:
For partner treatment, index women who were diagnosed with trichomonas vaginalis and index men who were diagnosed with urethritis were randomized to one of three study arms:

Standard partner referral (PR) - index patients were instructed to tell their partners that they need to go to a clinic for STI evaluation and treatment.

Booklet-enhanced partner referral (BEPR) - index patients were given a wallet-sized booklet containing 4 tear-out cards with information for the partner and treatment guidelines for the providers that would see the partners. The partners could then present this card at a clinic to help the clinician better treat them. If index patients had more than 4 partners, they were given additional booklets.

Patient delivered partner treatment (PDPT) - index patients were given packages containing 2 gram metronidazole (for TV patients) or azithromycin 1 gram and cefixime 400 mg (for urethritis patients) for up to 4 identified sex partners. When cefixime was no longer available, ciprofloxacin 500 mg was used. These packages contained written instructions about how to take the medication, warnings about side effects and a nurse's pager number to call if there were any questions or if the partner encountered any problems. All medications were distributed in containers with childproof caps and the partner's initial and birthdates were written on the bottle. This was a requirement of the Louisiana State Pharmacy Board. Names were not documented on the index patient's study or medical records.

ELIGIBILITY:
Inclusion Criteria:

* Woman attending Family Planning Clinic or men attending STD clinic
* Aged 16-44
* (non-pregnant women) - positive InPouch for trichomonas, or
* (pregnant women) - positive wet mount or InPouch for Trichomonas vaginalis
* (men) a complaint of urethritis which is verified on examination
* Report having >= 1sex partners in past 60 days
* Not presumptively treated for trichomonas (women) or urethritis (men)
* Provide informed consent to be re-contacted by telephone or in person in 14-28 days for a follow-up interview and T vaginalis or CT/GC rescreening

Exclusion Criteria:

Men

* Prisoner
* Has taken cefixime or azithromycin in last two weeks
* Has previously participated in the study
* All female partners are pregnant and did not have male partners Women
* client has taken metronidazole in the last two weeks
* client has been in this study previously
* women who are asymptomatic and in their first trimester of pregnancy

Ages: 16 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1500
Dates: Start 2001-12; Study Completion 2004-12

PRIMARY OUTCOMES:
Index patient report of partner taking medicine at 6-8 weeks

SECONDARY OUTCOMES:
Index patient re-infection at 6-8 weeks
Cost effectiveness outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Patty Kissinger, PhD, Principal Investigator — Tulane University School of Public Health and Tropical Medicine
Locations (2):
- United States (2):
  - Delgado STD Clinic, New Orleans, Louisiana
  - Orleans Women's Health Clinic, New Orleans, Louisiana

REFERENCES:
- [Result] Kissinger P, Mohammed H, Richardson-Alston G, Leichliter JS, Taylor SN, Martin DH, Farley TA. Patient-delivered partner treatment for male urethritis: a randomized, controlled trial. Clin Infect Dis. 2005 Sep 1;41(5):623-9. doi: 10.1086/432476. Epub 2005 Jul 19. PMID 16080084